CLINICAL TRIAL: NCT04780997
Title: The Effect of Virtual Reality Exercises on Balance in Patients With Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, MUSA POLAT, Asst.Prof.Dr, Nigde Omer Halisdemir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NigdeOHU
Record Dates: First submitted 2020-09-30; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Realty (Experimental): Microsoft Xbox Kinect® was used for virtual reality exercises
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Microsoft Xbox Kinect® was used for virtual reality exercises

SUMMARY:
Osteoporosis is a systemic disease characterized by low bone mass and increased bone fragility and increased fracture likelihood as a result of deterioration of the bone tissue microstructure.One of the important conditions determining the fracture risk in osteoporosis patients is fall. Balance exercises are perform to reduce the risk of falling.Virtual reality games are used in balance studies in many rehabilitation areas. The aim of this study is to investigate the effect of virtual reality exercises on balance.

DETAILED DESCRIPTION:
Osteoporosis is a systemic disease characterized by low bone mass and increased bone fragility and increased fracture likelihood as a result of deterioration of the bone tissue microstructure.One of the important conditions determining the fracture risk in osteoporosis patients is fall. Balance exercises are perform to reduce the risk of falling.Virtual reality games are used in balance studies in many rehabilitation areas. The aim of this study is to investigate the effect of virtual reality exercises on balance patients with osteoporozis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with primary osteoporosis

Exclusion Criteria:

* history of inflammatory rheumatic disease
* history of vestibular and cerebellar disease
* diseases affecting the central and peripheral nervous system (Parkinson's, stroke, ataxia, dementia, multiple sclerosis, peripheral neuropathy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Static balance index | 4th week
  Postural balance was measured using the Biodex Balance System (BBS) (Biodex Medical Systems, Shirley, NY), a movable balance platform that provides up to 20 of surface tilt in a 360 range of motion. The platform is interfaced with computer software (Biodex, Version 3.1, Biodex Medical Systems) that enables the device to serve as an objective assessment of balance

CONTACTS AND LOCATIONS:
Overall Officials: Musa Polat, Principal Investigator — Niğde OHÜ

IPD SHARING:
Plan to Share IPD: No